CLINICAL TRIAL: NCT00572000
Title: Safety Study of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) Vaccine in Healthy Vietnamese Women According to a 0, 1, 6 Month Schedule
Acronym: HPV-022 PRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute for Control of Vaccine and Biologicals (Other Government)
Responsible Party: National Institute for Control of Vaccine and Biologicals, National Institute for Control of Vaccine and Biologicals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111040 (HPV-022 PRI)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-10

CONDITIONS: Human Papillomavirus (HPV) Vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HPV-16/18 L1 VLP AS04 vaccine — Representation: 0.5ml monodose vials Administration: intramuscular Schedule: 0, 1, 6 month

SUMMARY:
The purpose of this study is to assess the occurrence of serious adverse events (SAEs) as well as evaluate the occurrence of solicited local and solicited general symptoms and the occurrence of medically significant conditions reported throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for vaccination visits and for the follow-up visit) should be enrolled in the study.

  • The female subject should be:
* married
* of Vietnamese origin, residing in Vietnam, and
* between, and including, 25 to 40 years of age at the time of the first vaccination.

  * Written informed consent obtained from the subject (prior to enrolment).
  * Healthy subjects as established by medical history and clinical examination before entering into the study.
  * Subjects must have a negative urine pregnancy test.
  * Subjects of childbearing potential (i.e. active menstrual cycle) at the time of study entry:
* must not be pregnant
* and must be abstinent (and if so, this must be documented in the source documents at each vaccination visit)
* or must be using adequate contraceptive precautions (i.e. intrauterine contraceptive device, oral contraceptives, diaphragm or condom in combination with contraceptive jelly, cream or foam, progestogen-only implantable cutaneous hormonal patch or injectable contraceptives) for 30 days prior to vaccination and must agree to continue such precautions for one month after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and up to one month after the last vaccine dose.

  * Subjects who have delivered recently or breastfeeding women must have completed a period of at least 3 months post-pregnancy and should not be breast-feeding in order to be enrolled in the study.

Planning to become pregnant or likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period.

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs on 14 consecutive days within six months prior to the first vaccine dose and up to one month after the last dose of the vaccine. (For corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before (Days - 1 to - 30) and 30 days (i.e. Days 0 - 29) after the first dose of vaccine. However, the administration of tetanus toxoid vaccine up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Any medically diagnosed or suspected immunodeficient condition such as human immunodeficiency virus (HIV) infection based on medical history and physical examination (no laboratory testing required).
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines, e.g. AS04, aluminium, MPL.
* Hypersensitivity to latex (found in syringe-tip cap and plunger).
* Known acute or chronic, clinically significant system conditions, e.g. neurologic,pulmonary, cardiovascular, hepatic, renal functional abnormality or psychiatric disorders, as determined by medical history, physical examination or previous laboratory tests.
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatic or kidney disease(s), diabetes, or autoimmune disease. This exclusion criterion should be understood as exclusion of subjects having significant medical conditions (such as cancer, autoimmune diseases) currently under treatment.
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Enrolment will be deferred until condition is resolved. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. oral/ axillary temperature < 37.5 °C (99.5 °F).
* A subject with body temperature (i.e. fever) > 37.5 °C (99.5 °F).
* Drug and/or alcohol abuse.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2007-11; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
To assess the occurrence of serious adverse events (SAEs) throughout the study | 7 months

SECONDARY OUTCOMES:
To evaluate the occurrence of solicited local and solicited general symptoms and the occurrence of unsolicited symptoms as well as the occurrence of medically significant conditions. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Son Hoa Hoang, Medicine Doctor, Principal Investigator — National Institute for Control of Vaccine and Biologicals
Locations (1):
- Thi Son commune health center and Ngoc Son Commune Health Center, Hà Nam, Vietnam